CLINICAL TRIAL: NCT05868486
Title: Whole Body MRI and Liquid Biopsy for Early Cancer Detection
Brief Title: Analysis of Whole Body Magnetic Resonance Imaging and Liquid Biopsy for Early Detection of Cancer in Patients With a Strong Family History of Cancer
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 21574; NCI-2022-01829 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 21574 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2023-03-29; First posted 2023-05-22 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Hematopoietic and Lymphoid System Neoplasm; Malignant Solid Neoplasm
MeSH Terms: interventions — Specimen Handling; Genetic Testing; Counseling; Liquid Biopsy; Contrast Media

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Whole Body MRI and Liquid Biopsy (Experimental): Patients undergo WBM without contrast and blood sample collection for liquid biopsy
  Interventions: Procedure: Biospecimen Collection; Genetic: Genetic Testing for Cancer Risk; Procedure: Liquid Biopsy; Procedure: Magnetic Resonance Imaging of the Whole Body without Contrast; Other: Survey Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Genetic: Genetic Testing for Cancer Risk — Undergo germline testing
  Other Names: Cancer Risk Assessment with Genetic Testing and Counseling
Procedure: Liquid Biopsy — Undergo liquid biopsy testing
  Other Names: Plasma Biopsy
Procedure: Magnetic Resonance Imaging of the Whole Body without Contrast — Undergo whole body MRI without contrast
  Other Names: WB-MRI without Contrast; Whole Body Magnetic Resonance Imaging without Contrast; Whole Body MRI without Contrast; Whole-body MRI without Contrast
Other: Survey Administration — Complete surveys

SUMMARY:
This study evaluates patient acceptability of whole body magnetic resonance imaging (WBM) and liquid biopsies (LB) in detecting early stage cancer in patients with a strong family history of cancer. Collecting family history and testing for genes passed on from parent to child (germline testing) can be used to predict the likelihood of a patient developing cancer. Currently, detection of early cancers focuses on screening specific organ systems such as breast and colon cancer. Magnetic resonance imaging (MRI) uses a large magnet and radio waves to look at organs and structures inside the body. Health care professionals use MRI scans to diagnose a variety of conditions, from torn ligaments to cancer. Liquid biopsy is test that analyzes blood samples to determine if cancer cells are present. This study may help researchers determine the feasibility of WBM and liquid biopsies to detect early stage cancer in patients that have a strong family history of cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the acceptability of the approach of LB and WBM.

SECONDARY OBJECTIVES:

I. Determine the prevalence of WBM findings requiring additional imaging or invasive testing.

II. Determine the effect of germline testing, LB, and WBM on psychological distress and health-related quality of life (HR-QOL) at 6 months after testing compared with baseline.

EXPLORATORY OBJECTIVE:

I. Determine correlation between high-risk LB findings and cancer detected on WBM.

OUTLINE: This is an observational study.

Patients undergo WBM without contrast, blood sample collection for liquid biopsy, and complete surveys on study. Germline testing may also be performed on blood sample collected as standard of care or using the Precision Medicine protocol (Institutional Review Board [IRB] 96144).

ELIGIBILITY:
Inclusion Criteria:

* Age >= 50 years, or age within 10 years of first degree relative with cancer at age of diagnosis (as long as age is >= 18)
* Have a strong family history of cancer ( >= 2 first-degree relatives with cancer, one first and second degree relative with cancer in one lineage (side of family), or at least three first or second degree relatives with cancer in one lineage (side of the family). Non-melanoma skin cancer excluded from family history eligibility
* Have a family history of early-onset cancer (age >40) in at least one first-degree relative
* Willing to have 50 mL of blood (approximately 3.5 tablespoons) drawn (40 ml if germline testing already performed)
* Able to undergo MRI (no implants, metal, or claustrophobia that would preclude MRI)
* Any cancer diagnosis within past 5 years, excluding non-melanoma skin cancer
* Positron emission tomography/computed tomography (PET/CT) or other whole body imaging modality (including combination of CT chest and abdomen) within 3 years
* No signs/symptoms of possible cancer (e.g. hemoptysis, breast mass, blood per rectum, unexplained weight loss)
* Willing to undergo standard of care genetic counseling and germline testing, or has already undergone genetic counseling and germline testing
* Documented informed consent of the participant

Exclusion Criteria:

* Unable to provide informed consent
* Contraindications to MRI (implants, metal, or claustrophobia that would preclude MRI)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-05-20 (Actual); Primary Completion 2026-10-19 (Estimated); Study Completion 2026-10-19 (Estimated)

PRIMARY OUTCOMES:
Acceptability of germline testing, liquid biopsy and whole body magnetic resonance imaging (WBM) | Up to 6 months after WBM
  Acceptability, as measured by the survey question "How satisfied are you with the research study overall?" and is defined as a score of 4 ("moderately acceptable) or 5 ("highly acceptable").

SECONDARY OUTCOMES:
Prevalence of WBM findings requiring additional imaging or invasive testing | Up to 6 months after WBM
  Prevalence of WBM findings requiring additional imaging or invasive testing, described as a per participant percentage.
Psychological distress (Germline testing)A | Up to 6 months after WBM
  The effect of germline testing on psychological distress, as measured by STAI survey composite score between baseline and 6 months after testing.
Psychological distress (Germline testing)B | Up to 6 months after WBM
  The effect of germline testing on psychological distress, as measured by cancer worry scale survey scores between baseline and 6 months after testing.
Psychological distress (Liquid Biopsy)A | Up to 6 months after WBM
  The effect of LB on psychological distress, as measured by STAI survey composite score between baseline and 6 months after testing.
Psychological distress (Liquid Biopsy)B | Up to 6 months after WBM
  The effect of LB on psychological distress, as measured by cancer worry scale survey scores between baseline and 6 months after testing.
Psychological distress (WBM)A | Up to 6 months after WBM
  The effect of Whole Body MRI on Psychological distress, as measured by STAI survey composite score between baseline and 6 months after testing.
Psychological distress (WBM)B | Up to 6 months after WBM
  The effect of Whole Body MRI on Psychological distress, as measured by cancer worry scale survey scores between baseline and 6 months after testing.
Health Related Quality of Life (HRQOL/Germline) | Up to 6 months after WBM
  The effect of germline testing on HRQOL, as measured by the change in SF12 survey composite score between baseline and 6 months after testing.
Health Related Quality of Life (HRQOL/LB) | Up to 6 months after WBM
  The effect of LB on HRQOL, as measured by the change in SF12 survey composite score between baseline and 6 months after testing.
Health Related Quality of Life (HRQOL/WBM) | Up to 6 months after WBM
  The effect of WBM on HRQOL, as measured by the change in SF12 survey composite score between baseline and 6 months after testing.

OTHER OUTCOMES:
Correlation between high-risk liquid biopsy findings and cancer detected on WBM | Up to 6 months after WBM
  Liquid biopsy (LB) test sensitivity and specificity calculated by comparing the LB results with the WBM results, with WBM results considered the gold standard. Confusion matrix statistics, such as positive predictive value, negative predictive value, and test accuracy examined. Results reported with their corresponding 95% confidence intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Dan Raz, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

REFERENCES:
- [Derived] Raz DJ, Nehoray B, Ceniceros A, Motarjem P, Landau S, Nelson RA, Gray SW. Feasibility of a cancer screening program using multicancer early detection testing and whole-body magnetic resonance imaging in a high-risk population. Cancer. 2025 Jan 1;131(1):e35709. doi: 10.1002/cncr.35709. PMID 39748640